CLINICAL TRIAL: NCT00719914
Title: IntraCoronary Treatment With Integrilin To Improve ANgiographic Outcomes (IC TITAN - TIMI 47) Trial
Brief Title: A Safety/Efficacy Study of Intracoronary Integrilin to Improve Balloon Angioplasty Outcomes for the Treatment of Heart Attacks
Acronym: IC TITAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, C. Michael Gibson, MS, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T101
Record Dates: First submitted 2008-01-07; First posted 2008-07-22 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-07

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: eptifibatide; Integrilin; ST-Elevation Myocardial Infarction; Acute Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Eptifibatide; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intracoronary injection of eptifibatide
  Interventions: Drug: eptifibatide
- 2 (Placebo Comparator): Intra-coronary injection of normal saline.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: eptifibatide — Intra-coronary injection, weight based, of eptifibatide.
  Arms: 1
Drug: eptifibatide — Intra-coronary injection, based on weight, of eptifibatide
  Arms: 1
Drug: normal saline — Intra-coronary injection, weight based, of normal saline.
  Arms: 2

SUMMARY:
The main purpose of this research study is to try to improve the results of the standard treatment for heart attacks. Normally, heart attack patients get a fast dose and a slow dose of eptifibatide in the emergency room, shortly after arriving. This drug is usually given through a vein in the arm. However, eptifibatide can also be injected directly into the heart's blood supply just before angioplasty, a common procedure to unblock a blood vessel in the heart. This new way of giving the drug is being studying.

DETAILED DESCRIPTION:
The primary objective of the IC-TITAN study is to demonstrate that an IC bolus of eptifibatide added to an upstream double-bolus and infusion regimen of eptifibatide administered intravenously and initiated early in the ER will result in significant additional clot resolution in vivo when compared with an IC injection of placebo (saline). The primary endpoint chosen to evaluate this hypothesis is the improvement in percent diameter stenosis of the culprit artery following the IC bolus administration of eptifibatide vs. IC placebo (saline) as assessed with quantitative coronary angiography (QCA).

ELIGIBILITY:
Inclusion Criteria:

Clinical

* Patients (men or women) at least 18 years of age and
* Presenting with ischemic chest discomfort >20 minutes and <6 hours of duration suggestive of acute myocardial infarction

AND:

ECG

* ST elevation >1mm (>0.1mV) in two contiguous limb leads OR >2mm (>0.2mV) in two contiguous precordial leads

Exclusion Criteria:

CLINICAL

* Maximal systolic blood pressure <80 mmHg AFTER initial fluid and/or pressor resuscitation
* Uncontrolled hypertension (SBP>180 OR DBP >110) at time of enrollment
* Ventricular fibrillation or ventricular tachycardia requiring DC cardioversion
* Sinus bradycardia (HR <50/min), third degree or advanced second degree heart block.
* Known pregnancy
* New or suspected new left bundle branch block

BIOCHEMICAL

* Known thrombocytopenia (platelet count <100,000)
* Known severe renal insufficiency (creatinine >4.0 mg/dL)

INCREASED BLEEDING RISK

* Active or recent (<1 year) bleeding or gastrointestinal hemorrhage
* Major surgery <1 month
* Known coagulopathy, platelet disorder or history of thrombocytopenia: If a patient is known to be on chronic warfarin therapy, the International Normalized Ratio (INR) must be known to be <1.6 in order for the patient to be included
* Known neoplasm
* Any history of hemorrhagic cerebrovascular disorder or active intracranial pathology

MEDICATIONS

* Administration of a fibrinolytic agent within 7 days
* Known allergy or contraindication to eptifibatide OR aspirin OR heparin
* Treatment with another GP IIb/IIIa inhibitor within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, M.D., Study Chair — The TIMI Study Group; C. Michael Gibson, M.D., Principal Investigator — The TIMI Study Group
Locations (3):
- United States (3):
  - Cardiology Research Associates, Ormond Beach, Florida
  - Crittenton Hospital Medical Center, Rochester, Michigan
  - Mid Ohio Heart Clinic, Mansfield, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Additional Bolus of Eptifibatide: Intracoronary injection of eptifibatide
- Bolus of Normal Saline: Intracoronary injection of normal saline.
Period: Overall Study
Arm/Group | Additional Bolus of Eptifibatide | Bolus of Normal Saline
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bolus of Normal Saline: Intra-coronary injection of normal saline.
- Total: Total of all reporting groups
Arm/Group | Additional Bolus of Eptifibatide | Bolus of Normal Saline | Total
Number analyzed (Participants) | 10 | 7 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.2) | 67 (9.5) | 61.6 (10.7)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 75 years | 9 | 6 | 15
  >=75 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Percent Diameter Stenosis of the Culprit Artery Following the IC Bolus Administration of Eptifibatide vs. IC Placebo (Saline) as Assessed With Quantitative Coronary Angiography (QCA)
Time Frame: 30 days
Population: study terminated due to low enrollment
Arm/Group | Additional Bolus of Eptifibatide | Bolus of Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Additional Bolus of Eptifibatide | Bolus of Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No